CLINICAL TRIAL: NCT00231491
Title: Efficacy and Safety of Botulinum Toxin A for the Treatment of Refractory Overactive Bladder (OAB). A Multicenter Phase II, Randomized, Double-blind, Placebo Controlled 6 Month Study . VESITOX
Brief Title: Efficacy and Safety of Botulinum Toxin A for the Treatment of Refractory Overactive Bladder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel OUSLIMANI, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P030438
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Urgency; Urge incontinence; Botulinum toxin A; Quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Botulinum Toxin A (Botox )

SUMMARY:
Overactive bladder induce urgency, urge incontinence, nocturia and pollakiuria. This condition is often resistant to anticholinergic drugs used as a first line treatment for this purpose. Moreover muscarinic side effects (constipation, mouth dryness) often limits the use of those treatments. This study is designed to evaluate the efficacy and safety of botulinum toxin A injected into the detrusor muscle to control symptoms and improve quality of life for patients resistant or intolerant to anticholinergic drugs.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of botulinum toxin A injected into the detrusor muscle to control symptoms and improve quality of life for patients resistant or intolerant to anticholinergic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder with more than 3 episodes of urgency of urge incontinence per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of urgency and urge incontinence episodes at 3 months after injection | at 3 months

SECONDARY OUTCOMES:
Number of micturition episodes on micturition chart per day | per day
Mean value of volume of urine per micturition
Mean delay between urgency and leakage Quality of life improvement by Iqol and EuroQol (EQ-5D)
Urodynamic parameters : Volume at first contraction, volume at first desire to void, volume at urgency, maximal bladder capacity, maximal detrusor pressure
Number of pads used per day
Number of patients with less than 3 episodes per day of leakages by urge incontinence or urgency per day
Residual volume of urine after flowmetry
Maximal flow
Visual analogic scale for pain for procedure
Biologic modifications
Ultrasound of kidneys
Toxin A antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DENYS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- RAYMOND POINCARE Hospital, Garches, France

REFERENCES:
- [Background] Rajkumar GN, Small DR, Mustafa AW, Conn G. A prospective study to evaluate the safety, tolerability, efficacy and durability of response of intravesical injection of botulinum toxin type A into detrusor muscle in patients with refractory idiopathic detrusor overactivity. BJU Int. 2005 Oct;96(6):848-52. doi: 10.1111/j.1464-410X.2005.05725.x. PMID 16153215
- [Derived] Denys P, Le Normand L, Ghout I, Costa P, Chartier-Kastler E, Grise P, Hermieu JF, Amarenco G, Karsenty G, Saussine C, Barbot F; VESITOX study group in France. Efficacy and safety of low doses of onabotulinumtoxinA for the treatment of refractory idiopathic overactive bladder: a multicentre, double-blind, randomised, placebo-controlled dose-ranging study. Eur Urol. 2012 Mar;61(3):520-9. doi: 10.1016/j.eururo.2011.10.028. Epub 2011 Oct 25. PMID 22036776